CLINICAL TRIAL: NCT02901912
Title: Effect of Diet and Exercise in the Gut Microbiota of Premenopausal Women:Correlation With Inflammatory and Oxidative Stress Parameters
Brief Title: Comparison of Gut Microbiota in Sedentary and Active Women
Status: Completed | Type: Observational
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Mar Larrosa, Principal investigator, Universidad Europea de Madrid
Other Study IDs: UEM0001
Record Dates: First submitted 2016-07-27; First posted 2016-09-15 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Sedentary
Keywords: physical activity; sedentarism; fecal enzymatic activity
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples With DNA — Bacterial DNA extracted from feces
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Active: Women who perform at least 3h of physical activity per week
- Sedentary: Women who did not perform any kind of exercise

SUMMARY:
Gut microbiota comparison of active and sedentary women

DETAILED DESCRIPTION:
Observational study comparing gut microbiota of people who did not practice any physical exercise (sedentary) with the gut microbiota of people who at least practice exercise a minimum of 3 hours per week but they were not professional athletes. Since the hormonal status and gender are factors that influence gut microbiota, this study has been conducted in premenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* healthy women

Exclusion Criteria:

* Smokers, pregnant, vegetarian, vegan, taking antibiotics in the last 3 months, any kind of disease, body mass index>25

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy women who do not perform exercise at all or practice at least 3 hours of exercise per week
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Physical activity | 7 days
  Physical activity was determined by accelerometry

SECONDARY OUTCOMES:
Gut microbiota | One year
  Gut microbiota determination by 16S rRNA Sequencing
Diet | 6 months
  Diet was determined with a food frequency questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Mar Larrosa, PhD, Principal Investigator — Universidad Europea de Madrid
Locations (1):
- Mar Larrosa, Villaviciosa de Odón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided